CLINICAL TRIAL: NCT02992431
Title: Participatory Patient Care Planning in Primary Care: Effectiveness and Feasibility in Patients With Hypertension, Ischemic Heart Disease or Diabetes
Brief Title: Participatory Patient Care Planning in Primary Care
Acronym: 4PHC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kuopio University Hospital (Other)
Collaborators: Siilinjärvi Health Center (Unknown); University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Pekka Mäntyselkä, Professor, Kuopio University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 749-1-2017
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Hypertension; Ischemic Heart Disease; Diabetes Mellitus
Keywords: patient care planning; primary health care; comorbidity
MeSH Terms: conditions — Hypertension; Myocardial Ischemia; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual care (Active Comparator): Usual care including standard disease specific follow-up with visit to general practitioner.
  Interventions: Other: Usual care
- Participatory patient care planning (Experimental): Intervention includes the patient activation questionnaire form, a visit to the nurse who conducts the measurements (blood pressure, waist measurement, weight and length) and a visit to the general practitioner who discusses and agrees with the patient about the treatment goals and follow-up resulting in the written PPCP.
  Interventions: Behavioral: Participatory patient care planning

INTERVENTIONS:
Behavioral: Participatory patient care planning — Intervention includes the patient activation questionnaire form, a visit to the nurse who conducts the measurements (blood pressure, waist measurement, weight and length) and a visit to the general practitioner who discusses and agrees with the patient about the treatment goals and follow-up resulting in the written PPCP.
  Arms: Participatory patient care planning
Other: Usual care — Usual care including standard disease specific follow-up with visit to general practitioner.
  Arms: Usual care

SUMMARY:
In the aging population, the prevalence of chronic diseases and multimorbidity has become common. Therefore, the planning and coordination of care have become more important. However, it is not known what kind of treatment plan should be and what kind of patients would benefit most of it.

This research focuses on the participatory patient care planning in primary health care. In general, the participatory patient care planning (PPCP) aims to engage patients in self-care, to improve the collaboration between patients and professionals and to improve the use of resources. The present study investigates the feasibility and effectiveness of the PPCP.

The specific research questions of the present study are: Does the PPCP have an impact on the patient's quality of life? Does the PPCP improve the quality of care in management of chronic diseases? Does the PPCP improve patient's commitment with self-care? Does the PPCP impact on the use of health care services? The data consists of people aged at least 18 years living in the municipality of Siilinjärvi with diabetes, coronary heart disease or hypertension and who are recorded in in Siilinjärvi Health Care Center electronic patient record. The participating patients are recruited from those who contacts SiiIinjärvi Health Care Center in order to have a follow-up visit because of the treatment of their disease. This study aims to recruit 700 patients.

The participants are allocated into the intervention group and into the control group receiving usual care. Intervention consists of the PPCP. This includes the patient activation questionnaire form, a visit to the nurse who conducts the measurements (blood pressure, waist measurement, weight and length) and a visit to the general practitioner who discusses and agrees with the patient about the treatment goals and follow-up resulting in the written PPCP.

The main out-come measures are the quality of health related life measured with the 15D; the level of patient's activity in self-care with the Patient Activation Measurement (PAM); life satisfaction, self-rated health, a reduction in productivity with the Work Productivity and Activity Impairment Questionnaire (WPAI: GH), and the disease specific measures (blood pressure, HbA1C, LDL-cholesterol, body mass index and waist measurement). In addition, pain intensity and interference (NRS 0-10), mood (BDI-21), the number of visits and phone calls and referrals are measured.

DETAILED DESCRIPTION:
This research focuses on the participatory patient care planning in primary health care. In general, the participatory patient care planning (PPCP) aims to engage patients in self-care, to improve the collaboration between patients and professionals and to improve the use of resources. The present study investigates the feasibility and effectiveness of the PPCP.

The specific research questions of the present study are: Does the PPCP have an impact on the patient's quality of life? Does the PPCP improve the quality of care in management of chronic diseases? Does the PPCP improve patient's commitment with self-care? Does the PPCP impact on the use of health care services? The data consists of people aged at least 18 years living in the municipality of Siilinjärvi with diabetes, coronary heart disease or hypertension and who are recorded in in Siilinjärvi Health Care Center electronic patient record. The participating patients are recruited from those who contacts SiiIinjärvi Health Care Center in order to have a follow-up visit because of the treatment of their disease. This study aims to recruit 700 patients.

The participants are allocated into the intervention group and into the control group receiving usual care. Intervention consists of the PPCP. This includes the patient activation questionnaire form, a visit to the nurse who conducts the measurements (blood pressure, waist measurement, weight and length) and a visit to the general practitioner who discusses and agrees with the patient about the treatment goals and follow-up resulting in the written PPCP.

The main out-come measures are the quality of health related life measured with the 15D; the level of patient's activity in self-care with the Patient Activation Measurement (PAM); life satisfaction, self-rated health, a reduction in productivity with the Work Productivity and Activity Impairment Questionnaire (WPAI: GH), and the disease specific measures (blood pressure, HbA1C, LDL-cholesterol, body mass index and waist measurement). In addition, pain intensity and interference (NRS 0-10), mood (BDI-21), the number of visits and phone calls and referrals are measured.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypertension, ischemic hearth disease or diabetes living in the municipality of Siilinjärvi

Exclusion Criteria:

* Permanent bed patient, terminal phase of any serious condition, severe decline in cognition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
15D | one year
  Health related quality of life

SECONDARY OUTCOMES:
WPAI | one year
  Work Productivity and Activity Impairment Questionnaire
PAM | one year
  Patient Activation Measurement
HbA1C | one year
  B -Hemoglobin-A1c
LDL | one year
  plasma LDL cholesterol
blood pressure | one year
  blood pressure
BMI | one year
  body mass index
waist measure | one year
  waist measure
visits to nurse | one year
  number of visits to nurse
visits to physician | one year
  number of visits to physician

CONTACTS AND LOCATIONS:
Overall Officials: Pekka T Mäntyselkä, Professor, Study Chair — University of Eastern Finland; Nina M Tusa, MD, Principal Investigator — University of Eastern Finland
Locations (1):
- Siilinjärvi Health Center, Siilinjärvi, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tusa N, Mikkonen U, Kautiainen H, Mantyselka P. Participatory care plan for primary care patients with long-term diseases: results after a 36-month follow-up of a randomized controlled trial. BMC Health Serv Res. 2025 Apr 12;25(1):536. doi: 10.1186/s12913-025-12660-6. PMID 40217248
- [Derived] Tusa N, Kautiainen H, Elfving P, Sinikallio S, Mantyselka P. Depressive symptoms decrease health-related quality of life of patients with coronary artery disease and diabetes: a 12-month follow up study in primary care. Scand J Prim Health Care. 2023 Sep;41(3):276-286. doi: 10.1080/02813432.2023.2233995. Epub 2023 Jul 16. PMID 37455531
- [Derived] Tusa N, Kautiainen H, Elfving P, Sinikallio S, Mantyselka P. Randomized controlled study of the impact of a participatory patient care plan among primary care patients with common chronic diseases: a one-year follow-up study. BMC Health Serv Res. 2021 Jul 20;21(1):715. doi: 10.1186/s12913-021-06716-6. PMID 34284783
- [Derived] Tusa N, Kautiainen H, Elfving P, Sinikallio S, Mantyselka P. Relationship between patient activation measurement and self-rated health in patients with chronic diseases. BMC Fam Pract. 2020 Nov 4;21(1):225. doi: 10.1186/s12875-020-01301-y. PMID 33148185